CLINICAL TRIAL: NCT01504334
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Trial for the Safety and Efficacy of Pirfenidone in the Treatment of Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Safety and Efficacy Study of Pirfenidone to Treat Idiopathic Pulmonary Fibrosis(IPF)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Kawin Technology Share-Holding Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Zuojun Xu, Chief Physician, Beijing Kawin Technology Share-Holding Co., Ltd.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KAWIN-001
Record Dates: First submitted 2011-12-30; First posted 2012-01-05 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — pirfenidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pirfenidone(200mg) (Experimental): Pirfenidone（200mg）tablets will be taken 3 times a day during the whole study process. For the first week, 1 tablet will be taken each time. For the second week, 2 tablets will be taken each time. From the third week to the 48th week, 3 tablets will be taken each time. Base drug Acetyl Cysteine Tablets（600mg）will be taken once a day, 1 tablet each time from the first to the 48th week.
  Interventions: Drug: Pirfenidone
- Placebo (without active ingredient) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pirfenidone — Pirfenidone（200mg）tablets will be taken 3 times a day during the whole study process. For the first week, 1 tablet will be taken each time. For the second week, 2 tablets will be taken each time. From the third week to the 48th week, 3 tablets will be taken each time. Base drug Acetyl Cysteine Tablets（600mg）will be taken once a day, 1 tablet each time from the first to the 48th week.
  Arms: Pirfenidone(200mg)
Drug: Placebo — Placebo（without active ingredient） tablets will be taken 3 times a day during the whole study process. For the first week, 1 tablet will be taken each time. For the second week, 2 tablets will be taken each time. From the third week to the 48th week, 3 tablets will be taken each time. Base drug Acetyl Cysteine Tablets（600mg）will be taken once a day, 1 tablet each time from the first to the 48th week for both groups.
  Arms: Placebo (without active ingredient)

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a chronic, progressive form of lung disease characterized by fibrosis of the supporting framework (interstitium) of the lungs. By definition, the term is used only when the cause of the pulmonary fibrosis is unknown ("idiopathic"). Microscopically, lung tissue from patients shows a characteristic set of histologic/pathologic features known as usual interstitial pneumonia (UIP). UIP is therefore the pathologic counterpart of IPF.Idiopathic pulmonary fibrosis is characterized by radiographically evident interstitial infiltrates predominantly affecting the lung bases and by progressive dyspnea and worsening of pulmonary function. No therapy has been clearly shown to prolong survival. The current strict definition of idiopathic pulmonary fibrosis provides a new focus for basic and clinical research that will improve insight into the pathogenesis of this disorder and stimulate the development of novel therapies.

Pirfenidone has proven antifibrotic and anti-inflammatory properties in various in vitro systems and animal models of pulmonary fibrosis, although its precise mechanism of action remains unclear. It attenuates fibroblast proliferation, production of fibrosis-associated proteins and cytokines, and the increased biosynthesis and accumulation of extracellular matrix in response to cytokines such as transforming growth factor-β. It is also shown to slow tumor cell proliferation by inhibiting fibroblast growth factor, epidermal growth factor and platelet-derived growth factor.

Pirfenidone has not been widely approved for clinical use in China, in this study, safety and efficacy were evaluated to see if pirfenidone has a significant advantage over placebo in terms of improving lung function and life quality etc. (see primary and secondary criteria) or slows down the deterioration of lung function in Chinese subjects diagnosed with IPF.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent signed;
2. 18-75 years of age;
3. Clinically or multidisciplinarily diagnosed idiopathic pulmonary fibrosis(see 2011 guidance );
4. Resting state PaO2≥50mg, FVC%≥45% normal predicted value and DLCO≥30% normal predicted value.

Exclusion Criteria:

1. Allergic to pirfenidone;
2. Dyspnea symptoms relieved in the past 6 months;
3. Patients in acute exacerbation phase;
4. Diabetic patients whose fasting venous glucose >11.1 mmol/L;
5. Patients with malignant tumor and hemorrhagic diseases;
6. Patients with serious underlying pulmonary disease;
7. Patients with serious heart disease(NYHA class Ⅲ-Ⅳ), liver disease(ALT or AST 2 times above the upper level of normal value range), kidney disease(Cr above the upper level of normal value range);
8. Patients who has taken Acetylcysteine in the past 3 months;
9. Patients who has taken Prednisone>15mg/day(or other equivalent amount of glucocorticoid) and/or Immunosuppresants in the past 3 months;
10. Patients who has taken interferon, penicillamine, colchine or other agents for the treatment of IPF;
11. Pregnant or lactating women;
12. Participated in other clinical trials in the past 1 month;
13. The investigator assessed as inappropriate to participate in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-11 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Changes in forced vital capacity (FVC) | 48 weeks
  Changes in FVC from 48 weeks to baseline

SECONDARY OUTCOMES:
Changes in lung function (including arterial blood gas analysis) | 48 weeks
  Lung function will be assessed as improved/stabilized/exacerbated from 48 weeks to baseline.
Acute Exacerbation during the whole treatment procedure（frequency and severity） | 48 weeks
  The following clinical deterioration symptoms within a month that cannot be explained by other reasons will be assessed as acute exacerbation:
  1. Aggravated dyspnea;
  2. Newly discovered chest interstitial lung abnormality by radiograph/HRCT, without pneumothorax or pleural effusion;
  3. PaO2 decreases ≥10mm Hg，heart failure or pulmonary embolism excluded.
  Acute Exacerbation can be assessed if 1 and 2 appear or 1 and 3 appear.
Progression-free time | 48 weeks
  Progression of disease during the whole study period is defined as follows:
  1. Progressive dyspnea (objective evaluation);
  2. FVC absolute value progressively and constantly decreases compared with baseline value;
  3. DLCO absolute value (after hemoglobin calibration) progressively and constantly decreases compared with baseline value;
  4. Fibrosis progressive deterioration by HRCT examination;
  5. Acute Exacerbation;
  6. Death caused by respiratory failure.
6 Minute Walk Test (6MWT )： Changes in 6 minute walk distance (6MWD) and SpO2 from 48 weeks to baseline | 48 weeks
  Method: The walking test is conducted in a corridor 33 meters long. The patient is instructed to "walk from end to end, covering as much ground as they can in the allotted time". The total distance ambulated in meters during the 6-minute walk test and the number of rest stops is recorded. 6MWD, weight, heart rate, BP, SpO2, and a self-reported rating of perceived exertion [modified Borg RPE scale rating (0 to 10 scale)] is recorded after the walk.
Borg RPE scale rating improvement rate during the whole study period | 48 weeks
  Patient percentage whose Borg RPE scale rating improves more than 1 level.
Lung interstitial change observed by HRCT | 48 weeks
  Changes in HRCT lung interstitial evaluation score from 48 weeks to baseline
Life quality: assessed by St. George respiratory questionnaire (SGRQ). | 48 weeks
  Life quality will be assessed as improved if SGRQ single or total score increased >4% when completing the trial; Life quality will be assessed as stabilized if SGRQ single or total score changes within the range of 4% when completing the trial; Life quality will be assessed as exacerbated if SGRQ single or total score decreased >4% when completing the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Zuojun, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijng, China

REFERENCES:
- [Derived] Huang H, Dai HP, Kang J, Chen BY, Sun TY, Xu ZJ. Double-Blind Randomized Trial of Pirfenidone in Chinese Idiopathic Pulmonary Fibrosis Patients. Medicine (Baltimore). 2015 Oct;94(42):e1600. doi: 10.1097/MD.0000000000001600. PMID 26496265